CLINICAL TRIAL: NCT00404079
Title: Phase 4 Study of Glucosamine Sulphate in the Treatment for Chronic Low Back Pain Patients With Degenerative Lumbar MRI Findings
Brief Title: The Glucosamine-study: The Effect of Glucosamine in Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Dr. Oliver Grundnes, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28130805
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-02

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucosamine Sulphate (Experimental)
  Interventions: Drug: Glucosamine sulphate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucosamine sulphate — Oral intake of 1500 mg glucosamine sulfate(from Pharma Nord) daily for 6 months
  Other Names: Glucosamine sulfata Pharma Nord
  Arms: Glucosamine Sulphate
Drug: Placebo — Oral intake of 3 placebo capsules (similiar looking to the glucosamine sulfate capsules)daily for 6 months
  Arms: Placebo

SUMMARY:
Low back pain (LBP) is the most frequent cause of sick leave and disability pension, and degenerative and osteoarthritic (OA) changes is a significant cause of pain and disability. Some indications exist for symptomatic and possible cartilage-structurmodifying effect on knee- and hip-osteoarthritis with glucosamine sulphate (GS). The OA process in the lumbar spine is most likely to OA processes in knees and hips, hence GS could have comparable symptomatic and structural effect on lumbar OA.

Study hypothesis: No difference in treatment effect exists between oral intake of GS- or placebo-capsules for patients' with chronic low back pain measured with Roland Morris Disability Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for more than 6 months
* Patient older than 25 years old
* MRI findings comparable with lumbar degenerative/osteoarthritic changes.

Exclusion Criteria:

* Spinal stenosis with neurological deficits
* Spinal prolapse with neurological deficits
* Rheumatoid arthritis, psoriatic arthritis,
* Old lumbar fractures
* Chronic pain syndromes (e.g. fibromyalgia)
* Psychosocial status not suitable for participation
* Pregnancy
* Breastfeeding
* Allergic to shellfish

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Grundnes, MD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ulleval Universtiy Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Wilkens P, Scheel IB, Grundnes O, Hellum C, Storheim K. Effect of glucosamine on pain-related disability in patients with chronic low back pain and degenerative lumbar osteoarthritis: a randomized controlled trial. JAMA. 2010 Jul 7;304(1):45-52. doi: 10.1001/jama.2010.893. PMID 20606148
- [Derived] Wilkens P, Storheim K, Scheel I, Berg L, Espeland A. No effect of 6-month intake of glucosamine sulfate on Modic changes or high intensity zones in the lumbar spine: sub-group analysis of a randomized controlled trial. J Negat Results Biomed. 2012 Aug 17;11:13. doi: 10.1186/1477-5751-11-13. PMID 22900984
- [Derived] Wilkens P, Scheel IB, Grundnes O, Hellum C, Storheim K. Prognostic factors of prolonged disability in patients with chronic low back pain and lumbar degeneration in primary care: a cohort study. Spine (Phila Pa 1976). 2013 Jan 1;38(1):65-74. doi: 10.1097/BRS.0b013e318263bb7b. PMID 22718223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at Oslo University Hospital Outpatient Clinic. Recruitment occurred between December 2006 and July 2008 in Oslo Norway, mostly via referrals by general practitioners, physiotherapists, and chiropractors.
Pre-assignment Details: Trial participation required no wash out, run-in or transtion phase. Patients were excluded if they fulfilled any of the exclusion criteria.
Groups:
- Glucosamine Sulphate: The glucosamine sulphate (1500 mg) was taken daily and oral in capsule forms for 6 months
- Placebo: Placebo was taken daily and orally in capsule forms for 6 months
Period: Overall Study
Arm/Group | Glucosamine Sulphate | Placebo
Started | 125 | 125
Completed | 103 | 105
Not Completed | 22 | 20
Not completed — Lost to follow up, adverse event etc | 22 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucosamine Sulphate | Placebo | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 115 | 228
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 67 | 121
  Male | 71 | 58 | 129
Region of Enrollment [Number; unit: participants]
  Norway | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Roland Morris Disability Questionnaire
Description: The primary outcome was scores on the Norwegian version of Roland Morris Disability Questionnaire (RMDQ). RMDQ is a widely used back-specific, self-administered measure of pain-related disability. Greater levels of disability give higher numbers on a 24-point scale. RMDQ has content and construct validity and internal consistency. It is also reproducible and sensitive to change over time for LBP patients. A 3-point reduction in the total RMDQ was a priori classified as a response to treatment.
Time Frame: 1 year
Population: The number of participants for analysis followed the intention to treat principle. Imputation was performed with mulitple imputation.
Measure: Mean (Standard Deviation); unit: units on a scale (0-24)
Groups:
- Placebo: Oral intake of placebo capsules
- Glucosamine Sulphate: Glucosamine sulphate was taken daily and orally in capsule forms for 6 months
Arm/Group | Placebo | Glucosamine Sulphate
Number analyzed (Participants) | 125 | 125
units on a scale (0-24) | 9 (4) | 9 (4)
Statistical Analysis 1: Comparison: Placebo; Null hypothesis was glucosamine sulfate is not superior to placebo to reduce pain and disability associated with chronic low back pain. Power calculation was based on a 3 point difference between the groups with the primary outcome. Data was analysed with linear mixed models; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Odds Ratio (OR) = 4.5, Standard Deviation 4
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Visual Analogue Scale
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: EuroQol-5D
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Reports of adverse events were collected during the intervention period of 6 months
Arm/Group | Glucosamine Sulphate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/125
Other Adverse Events (participants affected / at risk) | 0/125 | 0/125

LIMITATIONS AND CAVEATS:
Free participation and the focus on glucosamine may attract a certain type of patients with specific personality traits. Adjunctive management was permitted, which may influence outcome. Compliance was assessed by capsule counts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes